CLINICAL TRIAL: NCT01921296
Title: UMCC 2013.051: Prospective Pilot Study Evaluating the Use of Cyclobenzaprine for Treatment of Sleep Disturbance, Fatigue, and Musculoskeletal Symptoms in Aromatase Inhibitor-treated Breast Cancer Patients
Brief Title: Pilot Study of Cyclobenzaprine for Treatment of Sleep Disturbance in Aromatase Inhibitor-treated Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual terminated early because of poor accrual
Sponsor: Lynn Henry (Other)
Collaborators: Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Lynn Henry, Assistant Professor of Internal Med, University of Michigan Rogel Cancer Center
Organization: University of Michigan Rogel Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2013.051
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-03

CONDITIONS: Sleep Initiation and Maintenance Disorders; Pain
Keywords: Breast cancer; Aromatase inhibitor
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain; Breast Neoplasms | interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclobenzaprine (Experimental): Cyclobenzaprine (Flexeril) 5 milligrams orally 2 hours before bed, for a total of 24 weeks.
  Interventions: Drug: Cyclobenzaprine

INTERVENTIONS:
Drug: Cyclobenzaprine — 5 milligrams orally 2 hours before bedtime
  Other Names: Flexeril

SUMMARY:
Many women with breast cancer who are treated with aromatase inhibitor medications develop difficulty sleeping and fatigue during treatment. Some examples of aromatase inhibitor medications include anastrozole (Arimidex), exemestane (Aromasin), and letrozole (Femara). Frequently, sleeping pills do not work very well to improve sleep. Cyclobenzaprine (Flexeril) is a medication that was originally developed to treat muscle spasms. It may also improve sleep in patients with chronic pain disorders, such as fibromyalgia. In this study we are testing to see if cyclobenzaprine at bedtime will help improve sleep in women treated with aromatase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, age ≥ 18, postmenopausal.
* Histologically proven stage 0-III invasive carcinoma of the breast
* Initiating or have been receiving a standard dose of aromatase inhibitor therapy (letrozole 2.5mg once daily or exemestane 25mg once daily or anastrozole 1mg once daily) for up to a total of 48 months of AI therapy.
* Trouble sleeping during the past week. (After signing the informed consent document, subjects must also have a global PSQI score of ≥5)
* ECOG performance status 0-2 (see Appendix A).

Exclusion Criteria:

* Known hypersensitivity to cyclobenzaprine or any of the inactive ingredients
* Diagnosis of sleep apnea that is currently interfering with sleep or requiring CPAP, restless leg syndrome that is currently interfering with sleep or requiring medication, or Epworth sleepiness scale >10.
* Subjects with a history of hypothyroidism must have been on a stable dose of thyroid replacement medicine for at least 3 months prior to enrollment
* Treatment with steroids within 1 month
* Treatment with monoamine oxidase inhibitors (MAO-I) within 14 days of enrollment.
* Concurrent treatment with bupropion, MAO inhibitors, phenothiazines (including thioridazine), selegiline, tramadol, or medications known to prolong the QT interval (www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
* Currently primary psychiatric diagnosis (schizophrenia, psychosis) or suicidal ideation, history of bipolar disorder, or seizure disorder
* Known moderate or severe hepatic impairment
* History of congestive heart failure or cardiac arrhythmia (other than atrial fibrillation); myocardial infarction within the past 6 months
* Uncontrolled narrow-angle glaucoma
* Pregnant or breast feeding
* Serious or unstable medical condition that could likely lead to hospitalization during the course of the study or compromise study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclobenzaprine
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cyclobenzaprine
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 77.5 [77 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Experience an Improvement in Sleep Quality as Assessed Using the Pittsburgh Sleep Quality Index (PSQI) With 8 Weeks of Cyclobenzaprine Therapy.
Description: Will measure sleep quality using the Pittsburgh Sleep Quality Index at baseline and after 8 weeks of therapy with cyclobenzaprine. A total score is calculated for the Pittsburgh Sleep Quality Index. The total score ranges from 0-21, with higher scores representing worse sleep quality. Any reduction in PSQI total score was considered an improvement.
Time Frame: 8 weeks
Population: Only one of the two enrolled participants completed questionnaires after the baseline assessment
Measure: Number; unit: participant
Arm/Group | Cyclobenzaprine
Number analyzed (Participants) | 1
participant | 1

2. Secondary Outcome: Change in Fatigue Between Baseline and Week 8 With Cyclobenzaprine Therapy
Description: Will measure fatigue using the PROMIS fatigue questionnaire at baseline and after 8 weeks of therapy with cyclobenzaprine. The PROMIS Fatigue 7a score was calculated according to the information provided on the website. The raw score ranges from 7-35. The raw score is then converted to a T score according to the instruction on the website, with higher scores representing more fatigue. The T score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. The change in fatigue is calculated by subtracting the T score at baseline from the T score at 8 weeks. Positive values represent worsening of fatigue.
Time Frame: baseline and 8 weeks
Population: Only one of the two enrolled participants completed questionnaires after the baseline assessment
Measure: Mean (Full Range); unit: change in T score
Arm/Group | Cyclobenzaprine
Number analyzed (Participants) | 1
change in T score | 1.3 [1.3 to 1.3]

3. Secondary Outcome: Change in Average Pain Between Baseline and Week 8 With Cyclobenzaprine Therapy
Description: Will measure average pain using the Brief Pain Inventory at baseline and after 8 weeks of therapy with cyclobenzaprine. On the Brief Pain Inventory, average pain is reported using a 0-10 scale, with higher numbers reflecting more pain. Change is calculated by subtracting pain at baseline is from pain at 8 weeks. A positive value represents an increase in pain.
Time Frame: baseline and 8 weeks
Population: Only one of the two enrolled participants completed questionnaires after the baseline assessment
Measure: Mean (Full Range); unit: change in average pain
Arm/Group | Cyclobenzaprine
Number analyzed (Participants) | 1
change in average pain | -2 [-2 to -2]

4. Other Pre Specified Outcome: Percentage of Subjects Who Continue to Take Aromatase Inhibitor Therapy
Description: We will assess the number of patients who continue to take the original aromatase inhibitor medication at the 24 week timepoint, as assessed using patient self-report and medical records
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine
Number analyzed (Participants) | 2
percentage of participants | 100

5. Other Pre Specified Outcome: Percentage of Patients That Experience Adverse Events
Description: Persistence with cyclobenzaprine therapy for 24 weeks will be assessed using a medication diary. Safety will be assessed using CTCAE criteria
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Cyclobenzaprine
Number analyzed (Participants) | 2
percentage of participants | 100

ADVERSE EVENTS:
Arm/Group | Cyclobenzaprine
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclobenzaprine (N=2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Nervous System Disorder - Other (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was closed early for futility. The primary endpoint was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes